CLINICAL TRIAL: NCT00183014
Title: Trial to Increase Walking Among Sedentary Older Latinos
Brief Title: Caminemos! Trial to Increase Walking Among Sedentary Older Latinos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Catherine Sarkisian, MD, MSPH, UCLA Division of Geriatrics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0049; 5R01AG024460-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Aging; Sedentary Lifestyle
Keywords: behavior therapy; exercise; gait; physical activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): discussion session and exercise class
  Interventions: Behavioral: The Lifetime Fitness Program; Behavioral: Exercise class
- 2 (Active Comparator): exercise class only
  Interventions: Behavioral: Exercise class

INTERVENTIONS:
Behavioral: The Lifetime Fitness Program — A series of 4 weekly 1-hour group discussion sessions that utilize attribution retraining techniques from the field of motivational psychology in combination with behavioral strategies based in social cognitive theory; weekly for 4 weeks, monthly for 11 months, then every two months for 12 months (total duration = 24 months
  Arms: 1
Behavioral: Exercise class — 1-hour exercise class aimed at increasing strength, flexibility and endurance; weekly for 4 weeks, monthly for 11 months, then every two months for 12 months (total duration = 24 months

SUMMARY:
The purpose of this study is to examine the efficacy of a multifaceted behavioral intervention aimed at raising walking levels among sedentary older Latinos.

DETAILED DESCRIPTION:
Regular physical activity contributes to the health and quality of life of older adults, but unfortunately only 20% of men and 25% of women aged 65 years and greater meet the minimal national guidelines for physical activity. Older Latinos have higher rates of diseases that are most likely to benefit from physical activity, but have disproportionately high rates of sedentary lifestyle. To address this major public health problem, this study will implement and evaluate a multifaceted intervention to raise and sustain walking levels among older Latinos.

A total of 600 sedentary older Latinos will be recruited from community-based senior centers in the greater Los Angeles region. The specific aims of the study are to test the effect of the intervention on:

1. the change in steps per week measured by digital pedometer from baseline to 1, 12, and 24-month follow-up;
2. self-reported physical activity level and intervening constructs (including expectations regarding aging and self-efficacy expectations for physical activity);
3. psychosocial health constructs, physical performance measures, and clinical health outcomes.

The core of the intervention consists of a series of 4 weekly 1-hour group discussion sessions that utilize attribution retraining techniques from the field of motivational psychology in combination with behavioral strategies based in social cognitive theory. Discussion sessions will be conducted at senior centers and led by a bilingual health educator; each session will be followed by a 1-hour exercise class aimed at increasing strength, flexibility and endurance. During the discussion sessions, the health educator will administer a structured culturally-tailored curriculum in which participants are taught to raise their expectations for physical activity with aging and not to attribute being sedentary to "old age." The 4 weekly sessions will be followed by monthly sessions for 11 months, and sessions every 2 months for the following 12 months (total intervention duration = 24 months). Participants will be randomized to 1 of 2 arms:

1. intervention arm: receiving the discussion session and the exercise class;
2. control arm: receiving just the exercise class with the same frequency and duration as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Self-identifying as Latino/Hispanic
* Not currently participating in 20 minutes or more of physical activity 3 times a week
* Willingness to take brief physical activity screening test and if do not pass, provide the name of a physician who has seen the patient in the recent past

Exclusion Criteria:

* Plans to move from the area in the next 24 months
* Unable to participate in 1-hour group discussion
* Unable to walk
* Physician stating that patient is not medically able to participate
* Family member already participating
* Substantial cognitive impairment (determined by a screening test)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of steps per week on digital pedometer | baseline and 1, 12, and 24-months

SECONDARY OUTCOMES:
Self-reported physical activity level | baseline and 1, 12, and 24-months
beliefs about aging | baseline and 1, 12, and 24-months
self-efficacy | baseline and 1, 12, and 24-months
health-related quality of life | baseline and 1, 12, and 24-months
blood pressure | baseline and 1, 12, and 24-months
body mass index (BMI) | baseline and 1, 12, and 24-months
physical performance measures | baseline and 1, 12, and 24-months
hospital days | baseline and 1, 12, and 24-months
outpatient visits | baseline and 1, 12, and 24-months
restricted activity days | baseline and 1, 12, and 24-months
cognitive function | baseline and 1, 12, and 24-months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Sarkisian, MD, MSPH, Principal Investigator — UCLA Division of Geriatrics
Locations (1):
- UCLA Division of Geriatrics, Los Angeles, California, United States

REFERENCES:
- [Derived] Piedra LM, Andrade FCD, Hernandez R, Trejo L, Prohaska TR, Sarkisian CA. Let's walk! Age reattribution and physical activity among older Hispanic/Latino adults: results from the inverted exclamation markCaminemos! Randomized trial. BMC Public Health. 2018 Aug 3;18(1):964. doi: 10.1186/s12889-018-5850-6. PMID 30075709